CLINICAL TRIAL: NCT02098213
Title: Evaluation of Spa Therapy in the Treatment of Plaque Psoriasis, a Randomized, Controlled, Open Multicenter Study
Brief Title: Evaluation of Spa Therapy in the Treatment of Plaque Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association Francaise pour la Recherche Thermale (Other)
Collaborators: University Hospital, Grenoble (Other); Floralis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PSOTHERMES
Record Dates: First submitted 2014-03-17; First posted 2014-03-27 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Plaque Psoriasis
Keywords: plaque psoriasis; DLQI; VQ Dermato; PASI; PASI change; phototherapy; balneotherapy; hydrotherapy; Euroquol EQ 5d scale; Visual analogic scale; SPA treatment Scale; PSS

STUDY DESIGN:
Intervention Model Description: Taking into account the hypothesis of a proportion of patients with a DLQI≤10 (absence of repercussion or low impact of psoriasis on quality of life) of 25% at 4 months 1/2 in the arm immediate spa treatment versus 10% in the usual care group (late spa treatment), 113 patients per group is required, with an alpha 5% risk and a power of 80 %. Given the risk of potential patients lost to follow-up estimates of 15%, we plan to include 130 patients per randomisation group, so 260 patients in total.
  According to the protocol submitted to authorities, given the uncertainties of necessary hypothesis, a re-evaluation of the number of subjects required after the first 100 inclusions is planned. This reassessment will be carried out without intermediate analysis but in view of the results observed for the primary endpoint in mean and standard deviation (event driven).
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Spa treatment (Active Comparator): Three week course of spa treatment soon after randomization
  Interventions: Other: Immediate spa treatment
- Late Spa treatment (Sham Comparator): Three week course of spa treatment soon after 4,5 months visit
  Interventions: Other: Late Spa treatment

INTERVENTIONS:
Other: Immediate spa treatment — soon after randomization: Spa treatment of 3 weeks. Spa treatment : that best adapted to the concerned pathology and common to all participating of spa resorts (walk in a specially pool, whirlpool bath with automatic air and water massages cycles, massaging shower etc)
  Other Names: Spa treatment soon after randomisation
  Arms: Immediate Spa treatment
Other: Late Spa treatment — soon after 4,5 months visit: Spa treatment of 3 weeks. Spa treatment : that best adapted to the concerned pathology and common to all of spa resorts (walk in a specially pool, whirlpool bath with automatic air and water massages cycles, massaging shower etc)
  Other Names: Spa treatment after 4,5 months visit in the study
  Arms: Late Spa treatment

SUMMARY:
Assessment of quality of life after Spa therapy (4 ½ months follow-up) in the treatment of plaque psoriasis: Spa versus usual care in patients with plaque psoriasis.

DETAILED DESCRIPTION:
Psoriasis is one of the most common skin diseases, affecting 2-3% of the general population; more than 1 million people in France.

This auto-immune erythematosquamous inflammatory dermatosis occurs on a particular genetic background and has a chronic course. Psoriasis has a history as an indication for dermatological spa treatment (water cures in the Dead Sea). As these treatments are a combination of balneotherapy and heliotherapy, many recent studies have attempted to assess the value and position the relative benefit of each therapeutic element. Over the last four decades various different phototherapy techniques have been widely used in the treatment of psoriasis. The thermal option for many psoriasis patients depends on personal choice, or their doctor's or dermatologist's recommendation. In 1994 only one third of the 16,875 spa treatments for dermatological conditions (about 5625 cures) were for psoriasis, suggesting that spa treatment is underused as a treatment for psoriasis. Nobody can challenge the therapeutic contribution of biotherapy in the treatment of anatomically destructive diseases such as rheumatoid arthritis and psoriatic arthritis, but the use of these treatments is not without risk and economic impact. There is thus a need for less intensive treatments that have little risk of serious side effects and are less expensive.

The use of spa therapy in psoriasis should be understood as complementary and not an alternative to all other treatments. The choice of treatment is guided by the patient's characteristics and pathology (concomitant diseases, extent of lesions, treatment history) and the specialty (adverse effects, cumulative dose). In psoriasis it may be necessary to use different lines of treatment because psoriasis is a lifetime disease. Side effects of systemic treatments such as biotherapy, cyclosporine, methotrexate, synthetic retinoids, and also phototherapy (PUVA and UVB) are cumulative over time. A course of spa treatment should allow a respite before resorting to other systemic therapy.

However, the spa dermatology still suffers from a lack of large-scale evaluation and especially an objective assessment using reliable methodologies that limit bias. This is the purpose of this study.

There are no randomized controlled multicenter clinical trials evaluating spa treatment for psoriasis, although an Italian non-randomized study included a few dozen patients and confirmed the clinical benefit of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes, over 18 years of age, patients with plaque psoriasis for more than one year diagnosed by a dermatologist
* Stable treatment in the last 6 months
* DLQI score > 10
* patients volunteering for spa treatment within 6 weeks
* consenting to participate to the study with informed consent form signed after appropriate information
* Affiliation to the French social security system or equivalent

Exclusion Criteria:

* Pregnancy, parturient or breast feeding
* Psychiatric illness or social situation that would preclude study compliance
* Refusal of consent
* Refusal of spa treatment
* Contra-indication to spa treatment
* Phototherapy in the last 3 months
* Guttate, pustular or erythrodermic psoriasis Isolated nail psoriasis
* Spa therapy in the past year
* Person deprived of liberty or under legal guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Dermatology Quality of Life Index (DQLI) | 4 ½ months after randomisation
  proportion of patients with a score ≤ 10 at 4½ months in each arm of the study, spa treatment versus usual care.

SECONDARY OUTCOMES:
Specific Quality Of Life | 4 1/2, 6, 9 and 12 months after randomisation
  proportion of patients in each arm of the study (spa treatment versus usual care) for the following specific dermatology questionnaires : DLQI score ≤ 10 at 6, 9 and 12 months and VQ Dermato score > 35 at 4 1/2, 6, 9 and 12 months
Global Quality Of Life | 4 1/2, 6, 9 and 12 months after randomisation
  EuroQOL 5D questionnaire at 4 1/2, 6, 9 and 12 months
Clinical benefit of the psoriasis | 4 1/2, 6, 9 and 12 months after randomisation
  proportion of patients with a PASI (Psoriasis Area and Severity Index) 50 and PASI 75 at 4½, 6, 9 and 12 months in each arm of the study, spa treatment versus usual care.
pain and pruritus | 4 1/2, 6, 9 and 12 months after randomisation
  Self-administered questionnaire with Visual Analogue Scale for pain and for pruritus at 4 1/2, 6, 9, 12 months
Treatment follow up | 4 1/2, 6, 9 and 12 months after randomisation
  * Assessment of topical treatments within 12 months (number of tubes used per month)
  * Number of phototherapy sessions
  * Use of conventional systemic therapies (acitretin, methotrexate, cyclosporine) (number of weeks of treatment and dosage)
  * Number of weeks of treatment by biotherapy
  * Reduction in the use of the health care system (Number of hospitalizations and specialized consultations in connection with psoriasis or not) within 12 months
  * Reports on the use of complementary and alternative medicines within12 months
patient's examination | 4 1/2, 6, 9 and 12 months after randomisation
  Impact of the spa treatment on overall metabolism indicators in the year
  Will be collected at 4 1/2, 6, 9 and 12 months in the two groups:
  * height an weight (BMI calculation)
  * Waist measurement
  * Blood pressure
Safety evaluation | 4 1/2, 6, 9 and 12 months after randomisation
  Evaluation of all adverse events attributable to treatment, or not, according to the usual criteria of pharmacovigilance in clinical trials
Stress evaluation | 4 1/2, 6, 9 and 12 months after randomisatio
  self administered questionnaire (PSS: Assessment of stress) at inclusion in the study only
Long term evaluation | 12 months
  Evaluation of the maintenance of benefits at 12 months (stability of the long term effect) on the primary outcome and secondary outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Marie MB BEYLOT-BARRY, Professor, Principal Investigator — Bordeaux University Hospital - France
Locations (5):
- France (5):
  - Station Thermale Avene, Avène, Languedoc-Rousillon
  - Thermes de Molitg les bains, Molitg-les-Bains, Languedoc-Roussillon
  - Thermes La Roche Posay, La Roche-Posay, Poitou-Charentes
  - Les thermes de ST-GERVAIS, Le Fayet, Rhône-Alpe
  - Etablissement thermal d'Uriage, Uriage-les-Bains, Rhône-Alpe

REFERENCES:
- [Background] Halverstam CP, Lebwohl M. Nonstandard and off-label therapies for psoriasis. Clin Dermatol. 2008 Sep-Oct;26(5):546-53. doi: 10.1016/j.clindermatol.2007.10.023. PMID 18755374
- [Background] Kazandjieva J, Grozdev I, Darlenski R, Tsankov N. Climatotherapy of psoriasis. Clin Dermatol. 2008 Sep-Oct;26(5):477-85. doi: 10.1016/j.clindermatol.2008.05.001. PMID 18755366
- [Background] ALT J, NONCLERCQ E. [Treatment of psoriasis by ultraviolet and photosensitizers]. Bull Soc Fr Dermatol Syphiligr. 1953 Jul-Oct;60(4):343-5. No abstract available. Undetermined Language. PMID 13115903
- [Background] Grupper C, Bourgeois-Spinasse J, Eisenmann D. [Treatment of psoriasis in 1970]. Cah Med. 1970 Sep;11:Suppl:15-20. No abstract available. French. PMID 5454618
- [Background] Oddoze L, Temime P, Marchand JP, Benne M. [Combined oral meladinine and ultraviolet rays in the treatment of psoriasis. (Preliminary note)]. Bull Soc Fr Dermatol Syphiligr. 1967;74(5):609-10. No abstract available. French. PMID 5587899
- [Background] SOLOMON WM, NETHERTON EW, NELSON PA, ZEITER WJ. Treatment of psoriasis with Goeckerman technic. Arch Phys Med Rehabil. 1955 Feb;36(2):74-7. No abstract available. PMID 13229486
- [Background] Young E. Ultraviolet therapy of psoriasis: a critical study. Br J Dermatol. 1972 Oct;87(4):379-82. doi: 10.1111/j.1365-2133.1972.tb07426.x. No abstract available. PMID 4562168
- [Background] van de Kerkhof PC. Therapeutic strategies: rotational therapy and combinations. Clin Exp Dermatol. 2001 Jun;26(4):356-61. doi: 10.1046/j.1365-2230.2001.00829.x. PMID 11422189
- [Background] Weinstein GD, White GM. An approach to the treatment of moderate to severe psoriasis with rotational therapy. J Am Acad Dermatol. 1993 Mar;28(3):454-9. doi: 10.1016/0190-9622(93)70067-4. PMID 8445062
- [Background] Lebwohl M. Combining the new biologic agents with our current psoriasis armamentarium. J Am Acad Dermatol. 2003 Aug;49(2 Suppl):S118-24. doi: 10.1016/s0190-9622(03)01144-7. PMID 12894135
- [Background] Tabolli S, Calza A, Di Pietro C, Sampogna F, Abeni D. Quality of life of psoriasis patients before and after balneo -- or balneophototherapy. Yonsei Med J. 2009 Apr 30;50(2):215-21. doi: 10.3349/ymj.2009.50.2.215. PMID 19430554
- [Background] Grob JJ, Auquier P, Martin S, Lancon C, Bonerandi JJ. Development and validation of a quality of life measurement for chronic skin disorders in french: VQ-Dermato. The ReseaudEpidemiolo gie en Dermatologie. Dermatology. 1999;199(3):213-22. doi: 10.1159/000018250. PMID 10592400
- [Background] Hsu S, Papp KA, Lebwohl MG, Bagel J, Blauvelt A, Duffin KC, Crowley J, Eichenfield LF, Feldman SR, Fiorentino DF, Gelfand JM, Gottlieb AB, Jacobsen C, Kalb RE, Kavanaugh A, Korman NJ, Krueger GG, Michelon MA, Morison W, Ritchlin CT, Stein Gold L, Stone SP, Strober BE, Van Voorhees AS, Weiss SC, Wanat K, Bebo BF Jr; National Psoriasis Foundation Medical Board. Consensus guidelines for the management of plaque psoriasis. Arch Dermatol. 2012 Jan;148(1):95-102. doi: 10.1001/archdermatol.2011.1410. PMID 22250239
- [Background] Pathirana D, Ormerod AD, Saiag P, Smith C, Spuls PI, Nast A, Barker J, Bos JD, Burmester GR, Chimenti S, Dubertret L, Eberlein B, Erdmann R, Ferguson J, Girolomoni G, Gisondi P, Giunta A, Griffiths C, Honigsmann H, Hussain M, Jobling R, Karvonen SL, Kemeny L, Kopp I, Leonardi C, Maccarone M, Menter A, Mrowietz U, Naldi L, Nijsten T, Ortonne JP, Orzechowski HD, Rantanen T, Reich K, Reytan N, Richards H, Thio HB, van de Kerkhof P, Rzany B. European S3-guidelines on the systemic treatment of psoriasis vulgaris. J Eur Acad Dermatol Venereol. 2009 Oct;23 Suppl 2:1-70. doi: 10.1111/j.1468-3083.2009.03389.x. PMID 19712190
- [Background] Basra MK, Fenech R, Gatt RM, Salek MS, Finlay AY. The Dermatology Life Quality Index 1994-2007: a comprehensive review of validation data and clinical results. Br J Dermatol. 2008 Nov;159(5):997-1035. doi: 10.1111/j.1365-2133.2008.08832.x. Epub 2008 Sep 15. PMID 18795920
- [Background] Tsai TF, Ho JC, Song M, Szapary P, Guzzo C, Shen YK, Li S, Kim KJ, Kim TY, Choi JH, Youn JI; PEARL Investigators. Efficacy and safety of ustekinumab for the treatment of moderate-to-severe psoriasis: a phase III, randomized, placebo-controlled trial in Taiwanese and Korean patients (PEARL). J Dermatol Sci. 2011 Sep;63(3):154-63. doi: 10.1016/j.jdermsci.2011.05.005. Epub 2011 May 20. PMID 21741220
- [Background] Shikiar R, Bresnahan BW, Stone SP, Thompson C, Koo J, Revicki DA. Validity and reliability of patient reported outcomes used in psoriasis: results from two randomized clinical trials. Health Qual Life Outcomes. 2003 Oct 8;1:53. doi: 10.1186/1477-7525-1-53. PMID 14613569
- [Background] Shikiar R, Willian MK, Okun MM, Thompson CS, Revicki DA. The validity and responsiveness of three quality of life measures in the assessment of psoriasis patients: results of a phase II study. Health Qual Life Outcomes. 2006 Sep 27;4:71. doi: 10.1186/1477-7525-4-71. PMID 17005043
- [Background] Fredriksson T, Pettersson U. Severe psoriasis--oral therapy with a new retinoid. Dermatologica. 1978;157(4):238-44. doi: 10.1159/000250839. PMID 357213
- [Derived] Beylot-Barry M, Mahe E, Rolland C, de la Breteque MA, Eychenne C, Charles J, Payen C, Machet L, Vermorel C, Foote A, Roques C, Bosson JL. Evaluation of the benefit of thermal spa therapy in plaque psoriasis: the PSOTHERMES randomized clinical trial. Int J Biometeorol. 2022 Jun;66(6):1247-1256. doi: 10.1007/s00484-022-02273-7. Epub 2022 Mar 26. PMID 35347400